CLINICAL TRIAL: NCT07181772
Title: Evaluatıon of Trıage Education Gıven to Fırst And Emergency Aıd Students With a Vırtual Escape Room: A Randomızed Controlled Study
Brief Title: Virtual Escape Room Education and Triage
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Gülsüme Satir, Ass.Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-BİAEK/07-37; 12-2025-01-50 (Other Grant/Funding Number: Biruni Universty)
Record Dates: First submitted 2025-07-17; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Student Education
Keywords: learning; triage; virtual escape room

STUDY DESIGN:
Intervention Model Description: Data Collection from Experimental Group Students: Students in the experimental group, assigned according to randomization, will complete a Personal Information Form and a Triage Knowledge Scale via Google Forms. A Virtual Escape Room game will be played during the Triage Training. After the game, the Game Play Experience Scale will be administered, and the Triage Knowledge Scale will be administered one month after the training.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group trained with the Virtual Escape Room game (Experimental): Students in the experimental group will play a virtual escape room game.
  Interventions: Behavioral: virtual escape room
- The group trained with the power point (Active Comparator): Triage training will be given to students in the control group using the classical method of powerpoint presentation.
  Interventions: Behavioral: with Power point education

INTERVENTIONS:
Behavioral: virtual escape room — Triage training will be taught to students in the experimental group for the first time through a virtual escape room game.
  Arms: The group trained with the Virtual Escape Room game
Behavioral: with Power point education — The control group was trained using the traditional method using power point.
  Arms: The group trained with the power point

SUMMARY:
This study was planned as a randomized controlled experimental design to determine the effect of triage training given to First and Emergency Aid students via a virtual escape room.

This research aims to increase the triage knowledge of First and Emergency Aid students and to develop an alternative training method for healthcare professionals working in the prehospital field.

The research hypotheses are:

Hypothesis 0: Training provided to First and Emergency Aid students using a virtual escape room has no effect on triage knowledge.

Hypothesis 1: Training provided to First and Emergency Aid students using a virtual escape room has an effect on triage knowledge.

DETAILED DESCRIPTION:
The study participants were identified as 122 people using Gpower. Data will be collected using a Personal Information Form, the Triage Information Scale, the Virtual Escape Room in Triage Training, and the Gaming Experience Scale.

ELIGIBILITY:
Inclusion Criteria:

Emergency and first aid students Having a smartphone

Exclusion Criteria:

Not answering all the questions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-10-23 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Triage knowledge scale | 2 weeks
  The investigators expect the post-test score of the of the experimental group students to be higher than their pre-test score.
GAMEX | 2 weeks
  The investigators expect the training provided through the virtual escape room to result in higher scores on the GAMEX scale

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Increasing the decision once the work is completed
Supporting Information: Study Protocol
Time Frame: 3 months after the study ends
Access Criteria: with web

REFERENCES:
- [Background] Quek LH, Tan AJQ, Sim MJJ, Ignacio J, Harder N, Lamb A, Chua WL, Lau ST, Liaw SY. Educational escape rooms for healthcare students: A systematic review. Nurse Educ Today. 2024 Jan;132:106004. doi: 10.1016/j.nedt.2023.106004. Epub 2023 Oct 24. PMID 37924674
- [Background] Lopez-Belmonte J, Pozo-Sanchez S, Lampropoulos G, Moreno-Guerrero AJ. Design and validation of a questionnaire for the evaluation of educational experiences in the metaverse in Spanish students (METAEDU). Heliyon. 2022 Nov 2;8(11):e11364. doi: 10.1016/j.heliyon.2022.e11364. eCollection 2022 Nov. PMID 36387471
- [Background] Löffler, E., Schneider, B., Zanwar, T., & Asprion, P. M. (2021). Cysecescape 2.0-a virtual escape room to raise cybersecurity awareness. International Journal of Serious Games, 8(1), 59-70.
- Available data/document: virtual escape room link for students: gsatir@biruni.edu.tr — https://docs.google.com/forms/d/1IGzEsuxfcY0aDEJ5_3JbotdJqtI4fq0K5o06ETrlRm4/edit — virtual escape room for triage education